CLINICAL TRIAL: NCT05164367
Title: Single-Dose Pharmacokinetics of Atropine Oral Gel in Healthy Adults
Brief Title: Pharmacokinetics of Atropine Oral Gel
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Venkata Yellepeddi, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144918
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Sialorrhea
Keywords: Pharmacokinetics; Cerebral Palsy; Sialorrhea; Atropine sulfate gel
MeSH Terms: conditions — Cerebral Palsy; Sialorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.1 mg of atropine (Experimental): 1 gram of gel by topical application in the oral cavity once.
  Interventions: Drug: Atropine sulfate gel (0.01%)

INTERVENTIONS:
Drug: Atropine sulfate gel (0.01%) — A research nurse will measure 1 gram of gel using a calibrated measuring spoon and will provide it to the participant for self-administration.
  Other Names: Atropine gel, mucoadhesive atropine gel

SUMMARY:
To evaluate the single-dose pharmacokinetics of atropine gel formulation after topical administration in the oral cavity of healthy adults.

DETAILED DESCRIPTION:
This study is a single-dose, single-center, open-label study of the pharmacokinetics of atropine gel (0.01% w/w) after topical oral administration in healthy adults. Study participants will be recruited by Drs. Murphy, Darro, and Yellepeddi at the Center for Clinical and Translation Science (CCTS), University of Utah. Participants who meet eligibility criteria will be recruited in the study after signing informed consent. Each of the 10 participants will receive 1 gram of atropine gel (0.01% w/w) containing 0.1 mg atropine via self-administration of gel into the oral cavity. Dr. Yellepeddi is a licensed pharmacist in the State of Utah and will train subjects in the administration of atropine gel in the oral cavity. A series of timed blood samples (0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours, 7 mL each time point) will be collected in commercial tubes, and plasma will be separated by centrifugation. The plasma samples will be stored frozen until further analysis by the Center for Human Toxicology (CHT), University of Utah.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and authorization.
2. Study participants must be able to complete consent, and all study evaluations written in the English language.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing at the time of screening
2. Chemotherapy or radiotherapy treatment within the last three months
3. Severe renal impairment defined as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 calculated using the CKD-EPI creatinine equation:

   eGFR (mL/min/1.73 m2) = 141 x min(Scr/k, 1)α x max(Scr/k,1)-1.209 x 0.993Age x 1.018 [if female] x 1.159 [if black]

   Where,
   1. k=0.7 if female
   2. k=0.9 if male
   3. α=-0.329 if female
   4. α=-0.411 if male
   5. min=The minimum of Scr/k or 1
   6. max=The maximum of Scr/k or 1
   7. Scr = serum creatinine (mg/dL)
4. Acute hepatitis in the prior 6 months, a prior history of cirrhosis, acute hepatic failure, or acute decompensation of chronic hepatic failure; and/or any of the following blood test results, for any individual, when assessed for eligibility:

   1. Bilirubin > 3 x upper limit of normal (ULN). [ULN for bilirubin = 1.4 mg/dL]
   2. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 3 x ULN values used by the laboratory performing the test. [ULN for AST = 40 U/L, ULN for ALT = 60 U/L]
   3. Alkaline phosphatase (ALP) > 3 x ULN [ULN for ALP = 126 U/L)
5. Deforming lesions of the oral cavity
6. Previous head and/or neck radiotherapy
7. Patients with a history of hypersensitivity reaction towards atropine and/or Carbopol 980 NF or any carbomers
8. Patients with heart conditions such as congenital heart disease, heart failure, coronary heart disease, myocardial infarction, and arrhythmia
9. Patients with acute glaucoma that may be exacerbated with atropine administration.
10. Patients with partial pyloric stenosis or other diseases related to gastrointestinal obstruction.
11. Patients diagnosed with urinary retention
12. Treatment with any other investigational drug during the 30 days prior to enrollment into the study
13. Patients receiving anticholinergic medications at baseline.
14. Patients who are receiving immunosuppression
15. Patients who are actively being treated for an infection
16. Patients with a history of salivary gland obstruction or stones
17. Patients with a history of chronic lung disease or chronic obstructive pulmonary disease (COPD)
18. Patients with an artificial airway (tracheostomy)
19. Patient taking monoamine oxidase inhibitors

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluate pharmacokinetic parameter time to reach maximum plasma concentration (Tmax) in healthy adults to see if atropine will reach detectable concentrations in plasma following topical oral administration in gel formulation. | The Tmax will be evaluated at timepoints 0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours after administration of gel to the oral cavity.
  Calculate the pharmacokinetic parameter Tmax after topical oral administration of 0.01% atropine gel.
Evaluate pharmacokinetic parameter time to reach maximum plasma concentration (Cmax) in healthy adults to see if atropine will reach detectable concentrations in plasma following topical oral administration in gel formulation. | The Cmax will be evaluated at timepoints 0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours after administration of gel to the oral cavity.
  Calculate the pharmacokinetic parameter Cmax after topical oral administration of atropine gel
Evaluate pharmacokinetic parameter area under the curve (AUC) in healthy adults to see if atropine will reach detectable concentrations in plasma following topical oral administration in gel formulation. | The AUC will be evaluated at timepoints 0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours after administration of gel to the oral cavity.
  Calculate the pharmacokinetic parameter AUC after topical oral administration of atropine gel
Evaluate pharmacokinetic parameter volume of distribution (Vd) in healthy adults to see if atropine will reach detectable concentrations in plasma following topical oral administration in gel formulation. | The Vd will be evaluated at timepoints 0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours after administration of gel to the oral cavity.
  Calculate the pharmacokinetic parameter Vd after topical oral administration of atropine gel
Evaluate pharmacokinetic parameter clearance (CL) in healthy adults to see if atropine will reach detectable concentrations in plasma following topical oral administration in gel formulation. | The CL will be evaluated at timepoints 0, 5, 10, 15, 30, 60 minutes, and 2, 4, 6, 8, and 24 hours after administration of gel to the oral cavity.
  Calculate the pharmacokinetic parameter CL after topical oral administration of atropine gel

CONTACTS AND LOCATIONS:
Overall Officials: Venkata K. Yellepeddi, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid SM, Westbury C, Chong D, Johnstone BR, Guzys A, Reddihough DS. Long-term impact of saliva control surgery in children with disability. J Plast Reconstr Aesthet Surg. 2019 Jul;72(7):1193-1197. doi: 10.1016/j.bjps.2019.02.020. Epub 2019 Mar 2. PMID 30885525
- [Background] Speyer R, Cordier R, Kim JH, Cocks N, Michou E, Wilkes-Gillan S. Prevalence of drooling, swallowing, and feeding problems in cerebral palsy across the lifespan: a systematic review and meta-analyses. Dev Med Child Neurol. 2019 Nov;61(11):1249-1258. doi: 10.1111/dmcn.14316. Epub 2019 Jul 22. PMID 31328797
- [Background] Parkes J, Hill N, Platt MJ, Donnelly C. Oromotor dysfunction and communication impairments in children with cerebral palsy: a register study. Dev Med Child Neurol. 2010 Dec;52(12):1113-9. doi: 10.1111/j.1469-8749.2010.03765.x. Epub 2010 Aug 31. PMID 20813020
- [Background] Reid SM, McCutcheon J, Reddihough DS, Johnson H. Prevalence and predictors of drooling in 7- to 14-year-old children with cerebral palsy: a population study. Dev Med Child Neurol. 2012 Nov;54(11):1032-6. doi: 10.1111/j.1469-8749.2012.04382.x. Epub 2012 Aug 9. PMID 22881219
- [Background] Reid SM, Westbury C, Guzys AT, Reddihough DS. Anticholinergic medications for reducing drooling in children with developmental disability. Dev Med Child Neurol. 2020 Mar;62(3):346-353. doi: 10.1111/dmcn.14350. Epub 2019 Sep 8. PMID 31495925
- [Background] Norderyd J, Graf J, Marcusson A, Nilsson K, Sjostrand E, Steinwall G, Arleskog E, Bagesund M. Sublingual administration of atropine eyedrops in children with excessive drooling - a pilot study. Int J Paediatr Dent. 2017 Jan;27(1):22-29. doi: 10.1111/ipd.12219. Epub 2015 Dec 27. PMID 26708211
- [Background] Protus BM, Grauer PA, Kimbrel JM. Evaluation of atropine 1% ophthalmic solution administered sublingually for the management of terminal respiratory secretions. Am J Hosp Palliat Care. 2013 Jun;30(4):388-92. doi: 10.1177/1049909112453641. Epub 2012 Jul 24. PMID 22833553
- [Background] De Simone GG, Eisenchlas JH, Junin M, Pereyra F, Brizuela R. Atropine drops for drooling: a randomized controlled trial. Palliat Med. 2006 Oct;20(7):665-71. doi: 10.1177/0269216306071702. PMID 17060265
- [Background] Lawrence R, Bateman N. Surgical Management of the Drooling Child. Curr Otorhinolaryngol Rep. 2018;6(1):99-106. doi: 10.1007/s40136-018-0188-2. Epub 2018 Mar 20. PMID 29651363
- [Background] Leung JG, Schak KM. Potential problems surrounding the use of sublingually administered ophthalmic atropine for sialorrhea. Schizophr Res. 2017 Jul;185:202-203. doi: 10.1016/j.schres.2016.12.028. Epub 2016 Dec 30. No abstract available. PMID 28043733
- [Background] Singla AK, Chawla M, Singh A. Potential applications of carbomer in oral mucoadhesive controlled drug delivery system: a review. Drug Dev Ind Pharm. 2000 Sep;26(9):913-24. doi: 10.1081/ddc-100101318. PMID 10914315
- [Background] Keegan G, Smart J, Ingram M, Barnes L, Rees G, Burnett G. An in vitro assessment of bioadhesive zinc/carbomer complexes for antimicrobial therapy within the oral cavity. Int J Pharm. 2007 Aug 1;340(1-2):92-6. doi: 10.1016/j.ijpharm.2007.03.023. Epub 2007 Mar 24. PMID 17452085
- [Background] Kelly HM, Deasy PB, Busquet M, Torrance AA. Bioadhesive, rheological, lubricant and other aspects of an oral gel formulation intended for the treatment of xerostomia. Int J Pharm. 2004 Jul 8;278(2):391-406. doi: 10.1016/j.ijpharm.2004.03.022. PMID 15196643
- [Background] Allison RR, Ambrad AA, Arshoun Y, Carmel RJ, Ciuba DF, Feldman E, Finkelstein SE, Gandhavadi R, Heron DE, Lane SC, Longo JM, Meakin C, Papadopoulos D, Pruitt DE, Steinbrenner LM, Taylor MA, Wisbeck WM, Yuh GE, Nowotnik DP, Sonis ST. Multi-institutional, randomized, double-blind, placebo-controlled trial to assess the efficacy of a mucoadhesive hydrogel (MuGard) in mitigating oral mucositis symptoms in patients being treated with chemoradiation therapy for cancers of the head and neck. Cancer. 2014 May 1;120(9):1433-40. doi: 10.1002/cncr.28553. PMID 24877167
- [Background] Alcon (2018). Viscotears® Liquid Gel [carbomer (polyacrylic acid)] - Patient Information Leaflet
- [Background] Regulatory Information for Carbopol®* 971P NF Polymer & Carbopol® 71G NF Polymer. file:///C:/Users/u0840209/Downloads/TDS-328_Carbopol_971P_71G_Regulatory_PH_Version%20(1).pdf
- [Background] Zeller RS, Lee HM, Cavanaugh PF, Davidson J. Randomized Phase III evaluation of the efficacy and safety of a novel glycopyrrolate oral solution for the management of chronic severe drooling in children with cerebral palsy or other neurologic conditions. Ther Clin Risk Manag. 2012;8:15-23. doi: 10.2147/TCRM.S26893. Epub 2012 Jan 25. PMID 22298950
- [Background] Reid SM, Johnson HM, Reddihough DS. The Drooling Impact Scale: a measure of the impact of drooling in children with developmental disabilities. Dev Med Child Neurol. 2010 Feb;52(2):e23-8. doi: 10.1111/j.1469-8749.2009.03519.x. Epub 2009 Oct 15. PMID 19843155
- [Background] Jones JM, Watkins CA, Hand JS, Warren JJ, Cowen HJ. Comparison of three salivary flow rate assessment methods in an elderly population. Community Dent Oral Epidemiol. 2000 Jun;28(3):177-84. doi: 10.1034/j.1600-0528.2000.280303.x. PMID 10830644
- [Background] Navazesh M, Christensen CM. A comparison of whole mouth resting and stimulated salivary measurement procedures. J Dent Res. 1982 Oct;61(10):1158-62. doi: 10.1177/00220345820610100901. No abstract available. PMID 6956596
- [Background] Dias BLS, Fernandes AR, Maia HS Filho. Treatment of drooling with sublingual atropine sulfate in children and adolescents with cerebral palsy. Arq Neuropsiquiatr. 2017 May;75(5):282-287. doi: 10.1590/0004-282X20170033. PMID 28591387
- [Background] Azapagasi E, Kendirli T, Perk O, Kutluk G, Oz Tuncer G, Teber S, Cobanoglu N. Sublingual Atropine Sulfate Use for Sialorrhea in Pediatric Patients. J Pediatr Intensive Care. 2020 Sep;9(3):196-200. doi: 10.1055/s-0040-1708552. Epub 2020 Apr 7. PMID 32685247
- [Background] Rapoport A. Sublingual atropine drops for the treatment of pediatric sialorrhea. J Pain Symptom Manage. 2010 Nov;40(5):783-8. doi: 10.1016/j.jpainsymman.2010.02.007. Epub 2010 Jun 11. PMID 20541902
- See also: Prescribing information of Cuvposa-glycopyrrolate liquid. — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=d200bd44-9856-4104-a29e-a4cca3db6737